CLINICAL TRIAL: NCT05838976
Title: Validity and Reliability of the Shorter Version of the CTQ-SSS in Patients With Carpal Tunnel Syndrome: A Cross-sectional Study
Brief Title: Validity and Reliability of CTQ-SSS in Carpal Tunnel Syndrome.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: 012/00X0021
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Participants: This group will consist of at least 50 patients with carpal tunnel syndrome who are undergoing nonsurgical management. Participants will complete the shorter version of the CTQ-SSS and other functional measures, such as the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire and the Patient-Rated Wrist Evaluation (PRWE). The validity and reliability of the CTQ-SSS will be assessed in this group using test-retest reliability and internal consistency analyses, as well as construct validity analyses comparing CTQ-SSS scores with other functional measures.
  Interventions: Diagnostic Test: Shorter Version of the CTQ-SSS

INTERVENTIONS:
Diagnostic Test: Shorter Version of the CTQ-SSS — The intervention in this study is the administration of the shorter version of the CTQ-SSS, a validated questionnaire designed to assess the severity of symptoms and functional limitations associated with carpal tunnel syndrome. The CTQ-SSS consists of 8 items related to symptom severity and 2 items related to functional status. The scores for each set of items are combined to generate symptom severity and functional status scores, which will be used to assess the validity and reliability of the CTQ-SSS in patients with carpal tunnel syndrome undergoing nonsurgical management.

SUMMARY:
To determine the validity and reliability of the shorter version of the CTQ-SSS in patients with carpal tunnel syndrome (CTS) undergoing nonsurgical management.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with carpal tunnel syndrome based on clinical presentation and/or nerve conduction studies.
* Patients aged 18 years to 60 years old.
* Patients who are undergoing nonsurgical management for carpal tunnel syndrome.

Exclusion Criteria:

* Patients with a history of hand or wrist surgery within the past 6 months.
* Patients with severe hand or wrist pain that would prevent completion of the outcome measures or interfere with their ability to participate in the study.
* Patients with severe cognitive impairment or language barrier that would prevent understanding of the study instructions or interfere with their ability to participate in the study.
* Patients with any other medical condition that could affect hand function or interfere with test completion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of patients with carpal tunnel syndrome who are undergoing nonsurgical management.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Validity and Reliability of the Shorter Version of the CTQ-SSS | Outcome measures will be assessed within 2-4 weeks of the initial CTQ-SSS administration.
  To determine the validity and reliability of the shorter version of the CTQ-SSS in patients with carpal tunnel syndrome undergoing nonsurgical management. The CTQ-SSS will be administered at baseline and at a follow-up visit within 2-4 weeks to assess test-retest reliability. Internal consistency will be assessed using Cronbach's alpha coefficient. Construct validity will be assessed by comparing the CTQ-SSS scores with other functional measures such as the DASH questionnaire and PRWE using Pearson's correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) collected during this study will be available upon reasonable request. Requests for access to the data should be submitted via email to mohamed.elmeligie@acu.edu.eg. All requests will be reviewed by the study investigators to ensure that they are reasonable and consistent with the ethical principles of the study. Access to the data will be granted in compliance with applicable laws and regulations, and with appropriate safeguards to protect the privacy and confidentiality of study participants.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: During the trial and after the trial by 6 months
Access Criteria: via email to mohamed.elmeligie@acu.edu.eg